CLINICAL TRIAL: NCT06328439
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ANS014004 Monotherapy in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate ANS014004 in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other); Hunan Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Zhejiang Cancer Hospital (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANS014004-I-CN-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: Part 1:
  QD: 7.5mg, 15 mg, 30 mg, 45 mg, 60 mg, 75mg, 90mg, 105mg, 120mg or 7.5mg, 15 mg, 22.5mg, 37.5mg, 52.5mg, 67.5mg BID: 30mg, 37.5mg, 45mg, 52.5mg, 60mg
  Part 2:
  RP2D as specified in Part 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANS014004 (Experimental): Dosage: 1. Dose-escalation participants receive ANS014004 single dose on Day 1, if DLT does not occur within the 3-day elution period, subjects will begin multiple doses on Day 8 and receive ANS014004 QD/BID for a 28-day cycle. 2, Backfill, Dose Extension Subjects, who go directly to multiple dosing, will receive ANS014004 QD/BID for 28 days as a cycle.
  Dosing Schedule: 1. Dose-escalation subjects, single dosing + multiple dosing, 31-day cycle. 2, Backfill, dose-expansion subjects, direct access to multiple dosing, 28 days to a cycle.
  Interventions: Drug: ANS014004

INTERVENTIONS:
Drug: ANS014004 — Specification: 7.5mg; 30mg QD/BID Oral

SUMMARY:
Brief Summary: This is a Phase I, first-in-human, open-label, multi-center study designed to explore the safety, tolerability, PK, and anti-tumor antitumor activity of ANS014004 monotherapy in subjects with locally advanced or metastatic solid tumors.

* The study consists of two parts: a dose-escalation part (Part 1) and a dose-expansion part (Part 2). For each subject, the study will consist of a screening period (Day -28 to Day -1), a treatment period (until discontinuation of treatment) and a follow-up period (including safety follow-up and survival follow-up).
* During the Treatment Period, subjects will receive ANS014004 single-agent oral administration until the subject meets any treatment termination criteria.

  1. The dose escalation phase (Part 1) will consist of a single-dose period and a multiple-dose period (28 days as one cycle). Subjects in the dose escalation phase will receive a single dose of ANS014004 on Day 1 of the single-dose period to obtain the complete PK profile of a single dose. There will be a 7-day washout period between the single-dose period and the multiple-dose period at the same dose level. If no dose-limiting toxicity (DLT) occurs within the 7-day washout period, subjects will start multiple-dose treatment on Day 8 (28 days per cycle), receiving ANS014004 once daily (QD) or twice daily (BID). Dose escalation will first be conducted in the QD dosing cohort. When the dose escalates to Cohort 5, dose escalation in the BID dosing cohort with the same daily dose will be conducted in parallel. For each group with the same daily dose of QD or BID cohorts, subjects will be enrolled in the QD cohort first, followed by the BID cohort, and then dose escalation of the next daily dose of QD or BID cohorts will be conducted. Both the QD and BID dosing cohorts will include a single-dose period and a multiple-dose period. Based on the safety, PK and preliminary efficacy data of the QD and BID cohorts, the dosing frequency and dose of the backfill cohort will be selected. Subjects in the backfill cohort will directly enter the multiple-dose period. The RP2D will be determined based on the comprehensive assessment of safety, PK and preliminary efficacy data from the dose escalation phase.
  2. In the dose expansion portion (Part 2), subjects will receive oral administration of ANS014004 at the RP2D dose QD or BID in each treatment cycle (28 days per cycle). The end-of-treatment (EOT) visit will be conducted within 7 days after the last dose or when the investigator decides to discontinue treatment. During the study period, the investigator and the sponsor may discuss and decide whether to stop exploring certain dose cohorts or to add exploration of other doses or dosing regimens based on the safety, PK and preliminary efficacy data obtained previously.

All subjects will undergo imaging evaluations of their tumors every 8 weeks until disease progression is confirmed by the investigator, the subject begins new antitumor therapy, dies, is lost to follow-up, or withdraws from the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ≥18 years of age at the time of signing the informed consent form.
2. Participants with a histologically confirmed diagnosis of unresectable locally advanced or metastatic solid tumors, relapsed or refractory to existing standard therapy, intolerant or unsuitable for existing standard therapy, or for whom no standard therapy is available (standard therapy is defined as therapy recommended by established guidelines and consensus [including, but not limited to, chemotherapy, radiotherapy, targeted therapy based on mutation status, immunotherapy, and surgery]). Locally advanced participants must be ineligible for radical surgery or radiotherapy. Participants who are intolerant of or unsuitable for existing standard therapy or for whom no standard therapy is available will be required to document these reasons.
3. Documentary evidence of pathogenic MET alterations from a local laboratory accredited by the Clinical Laboratory Improvement Act Amendments (CLIA), the International Organization for Standardization/Independent Ethics Committee (ISO/IEC), the College of American Pathologists (CAP), or other equivalent accreditation. Part 1 Specific Inclusion Criteria: Subjects carrying pathogenic MET alterations (including MET mutations, MET amplification, MET overexpression, MET fusions) will be enrolled. Part 2 Specific Inclusion Criteria: Subjects will be enrolled into one of the following 5 cohorts based on tumor type, MET alteration status, and prior therapy. Cohort 1: Subjects must have pathologically confirmed, diagnosed NSCLC with a MET exon 14 jump mutation, with or without other MET alterations, and prior treatment with an approved MET-TKI (e.g., camatinib and topotecanib). Cohort 2: Subjects must have pathologically confirmed, diagnosed NSCLC with a MET exon 14 jump mutation, with or without other MET alterations, relapsed or refractory to platinum-based chemotherapy, or intolerant or unsuitable for platinum-based chemotherapy, and have not received a prior MET-TKI. Cohort 3: Subjects must have pathologically confirmed, diagnosed NSCLC with a MET amplification, no MET exon 14 jump mutation, relapsed or refractory to platinum-based agent chemotherapy, intolerant to platinum-based agent chemotherapy, or unsuitable for platinum-based agent chemotherapy. Cohort 4: Subjects must have pathologically confirmed, diagnosed solid tumors (other than NSCLC) with MET exon 14 jump mutations, with or without other MET alterations, relapsed or refractory to standard therapy, or intolerant or unsuitable for standard therapy, or no standard therapy available. Cohort 5: Subjects must have a pathologically confirmed, diagnosed solid tumor with MET amplification (except NSCLC) or overexpression or fusion, without MET exon 14 jump mutations, relapsed or refractory to standard therapy, or intolerant or unsuitable for standard therapy, or no standard therapy available.
4. At least one measurable target lesion as defined by RECIST v1.1 (Appendix 3). (except for the low dose groups 7.5mg and 15mg).
5. Part 1 ECOG PS ≤ 1; Part 2 ECOG PS ≤ 2.
6. expected survival of ≥ 12 weeks in the judgment of the investigator.
7. Good organ function as determined by medical evaluation (within 7 days prior to study treatment), including: Good hematologic status, defined as: absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L, hemoglobin ≥ 90 g/L, and platelets ≥ 75 x 109/L. Receipt of platelet transfusions is not permitted within 3 days prior to testing, erythrocyte transfusions within 14 days prior to testing, and hematopoietic growth factors (polyethylene glycolized granulocyte colony-stimulating factor [G-CSF] or erythropoietin is within 14 days prior to testing) within 7 days prior to testing. Hematopoietic growth factors (polyethylene glycolated granulocyte colony-stimulating factor [G-CSF] or erythropoietin for up to 14 days prior to testing) are not allowed within days. Good hepatic function, defined as serum TBIL ≤ 1.5 x ULN (TBIL ≤ 3 x ULN with direct bilirubin ≤ 1.5 x ULN in subjects known to have Gilbert's syndrome), and serum ALT or AST ≤ 2.5 x ULN (or 5.0 x ULN in subjects with confirmed liver metastases). Good renal function, defined as creatinine clearance ≥ 50 mL/min (measured or calculated by the Cockcroft-Gault formula [Appendix 4]). Good coagulation function, defined as (including when receiving anticoagulation): prothrombin time (PT) < 1.5 x ULN and activated partial thromboplastin time (APTT) < 1.5 x ULN If subjects are receiving anticoagulation, they must have received a stable dose of anticoagulant for at least 1 month prior to study treatment.
8. Female subjects should use adequate contraception until 90 days after EOT, should not be breastfeeding, and must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test within 7 days prior to initiation of dosing for female subjects of childbearing potential; female subjects of childless potential must meet one of the following criteria at screening: Postmenopausal defined as amenorrhea for at least 12 months after cessation of all exogenous hormone therapy (if applicable). applicable) followed by amenorrhea for at least 12 months. Irreversible surgical sterilization such as hysterectomy, bilateral salpingo-oophorectomy, or bilateral salpingo-oophorectomy (as opposed to tubal ligation) has been clearly documented.
9. Male subjects whose female partners are of childbearing potential are required to use adequate contraception (i.e., barrier methods) during study participation and for 90 days after EOT. Male subjects must also refrain from sperm donation during study participation and for 90 days after the last dose of study treatment.
10. Be able to provide signed informed consent and comply with the requirements and limitations outlined in the Informed Consent Form (ICF) and in this study.

Exclusion Criteria:

1. for dose extension only (Part 2): known major driver gene alterations other than MET. For example, NSCLC harboring targeted alterations such as EGFR, ALK, RET, ROS1, BRAF, KRAS, etc. Investigators should discuss enrollment with sponsors regarding co-mutations.
2. Prior treatment with other type II MET-TKIs such as cabozantinib, glitinib, and melatinib (type II MET-TKIs are multi-targeted inhibitors that bind to the inactive conformation (DFG-out) of MET in the ATP pocket).
3. Participation in another therapeutic clinical trial within 28 days prior to the first study dose.
4. Received antineoplastic therapy (chemotherapy, immunotherapy, hormone therapy, targeted therapy, biologic therapy, or other antineoplastic therapy, except for hypothyroid hormone or estrogen replacement therapy, anti-estrogen analogs, or agonists required for suppression of serum testosterone levels) within 14 days or 5 half-lives (whichever is shorter) of the first dose of study treatment. The following exceptions apply: 1) Received nitrosourea or mitomycin C within 6 weeks prior to the first dose of study treatment. 2) Received a proprietary medicine with an antitumor indication within 7 days prior to the first dose of study treatment.
5. has received wide-field radiotherapy within 28 days prior to the first dose of study treatment or has received palliative localized radiotherapy within 14 days prior to the first dose of study treatment. Subjects must have recovered from all radiotherapy-related toxicities and not require corticosteroids.
6. Underwent major surgery (excluding diagnostic procedures) within 4 weeks prior to the initial study treatment, or is expected to require major surgery during the study period.
7. Toxicity from prior therapy has not subsided to ≤ Grade 1 or baseline levels as evaluated by NCI-CTCAE v5.0. Note: For certain Grade 2 toxicities (e.g., alopecia, skin pigmentation, neuropathy), subjects may be enrolled if the toxicity is stable and does not compromise the safety of participation in this study.
8. History of another primary solid tumor diagnosed or requiring treatment within the past 3 years (with the exception of localized basal cell or squamous cell carcinoma of the skin that has been adequately treated; or any other carcinoma in situ currently in complete remission).
9. Presence of CNS metastases that are known to be symptomatic or clinically unstable or that require an increased steroid dose to manage central nervous system (CNS) symptoms within 4 weeks prior to the first study dose. Note: Subjects with symptomatic CNS metastases may be enrolled in the study after treatment and control of their symptoms provided they have been clinically stable for at least 2 weeks, have no evidence of new brain metastases or enlargement of brain metastases, and have not had an increase in steroid dose to manage CNS symptoms within 4 weeks prior to the first study dose. Persons with comorbid carcinomatous meningitis or meningeal spread or spinal cord compression were not eligible for enrollment, regardless of whether they were clinically stable.
10. The subject is receiving an unstable or escalating dose of corticosteroids. For subjects receiving corticosteroids for endocrine defects or disease-related symptoms (excluding CNS disease), the dose must have been stabilized (or lowered) for at least 14 days prior to the first dose of study treatment.
11. the presence of any evidence of severe or uncontrolled systemic disease, as judged by the investigator, including, but not limited to: uncontrolled hypertension, defined as a systolic blood pressure (BP) ≥160 mmHg or diastolic BP ≥100 mmHg despite medication. for subjects with a history of hypertension, enrollment is permitted if the BP is stable and is controlled within these limits with antihypertensive therapy. Prior history of, or current clinical symptoms of, interstitial lung disease or interstitial pneumonia, or high risk of interstitial lung disease or interstitial pneumonia, including radiation pneumonitis (i.e., interfering with activities of daily living or requiring therapeutic intervention). Unstable or decompensated respiratory and renal disease, active bleeding disorders.
12. Serious cardiovascular or cerebrovascular disease including, but not limited to: Mean Fridericia formula-corrected QT intervals (QTcF) > 470 ms obtained on three repetitions of 12-lead electrocardiograms (ECGs) at rest Symptomatic heart failure with a New York Heart Association (NYHA) cardiac function classification of class II or higher. Echocardiographic (ECHO) assessment showing a baseline left ventricular ejection fraction (LVEF) below the lower limit of institutional normal (LLN) or < 50%. Any clinically significant rhythmic, conduction, or morphologic abnormality as demonstrated by resting ECG results, e.g., complete left bundle branch block, third-degree heart block, ventricular arrhythmia requiring antiarrhythmic therapy. Any of the following within 6 months prior to the first dose of study treatment: myocardial infarction, severe/unstable angina, coronary artery bypass grafting, congestive heart failure, cardiomyopathy, pulmonary embolism, cerebral vascular accident, or transient ischemic attack.
13. Presence of uncontrolled co-infections including, but not limited to: active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. If hepatitis B surface antigen (HBsAg) positive, HBV DNA testing should be performed. Subjects may be eligible to participate in the study if HBV DNA is <500 IU/ml or if the test value is below the lower limit of detection at the study center. (Subjects with primary liver cancer may be eligible for enrollment if HBV DNA <2000IU/ml) If HCV antibody is positive, HCV ribonucleic acid (RNA) testing should be performed. If HCV RNA is negative, the subject may be eligible for the study. Known human immunodeficiency virus (HIV) infection or known history of acquired immunodeficiency syndrome (AIDS), HIV positive. Active tuberculosis infection. Active infection requiring systemic therapy that occurred within 14 days prior to the first dose of study treatment.
14. Unwillingness or inability to comply with oral drug administration requirements or the presence of gastrointestinal disorders such as refractory nausea and vomiting, any acute or chronic gastrointestinal disorder, inability to swallow preparations, or previous major colectomy may prevent adequate absorption of ANS014004.
15. Concomitant use of drugs metabolized by P-glycoprotein (P-gp)/Breast cancer resistance protein (BCRP) or OCT2/OATP1B1/MATE1 within five half-lives prior to the administration of study therapy, or treatment with potent inducers or inhibitors of CYP2B6, CYP2C9, CYP2C19, OCT2, OATP1B1, or MATE1. For dose escalation only: Treatment with moderate or strong inducers or inhibitors of CYP2C8, CYP2D6, or CYP3A4 during the five half-lives preceding the administration of study therapy.
16. Combined use of acid-regulating drugs (e.g., proton pump inhibitors [PPIs] and H2 blockers) within 5 half-lives prior to use of study treatment.
17. Presence of pleural effusion, pericardial effusion or ascites requiring drainage and/or causing severe clinical symptoms (e.g., causing shortness of breath, tachycardia, etc.).
18. Previous or ongoing severe retinopathy.
19. History of allergic reaction to ANS014004 or its excipients, or to drugs with a similar chemical or biological structure or class to ANS014004.
20. received any live attenuated vaccination within 30 days prior to the first dose of study treatment.
21. known to have a psychiatric or substance abuse disorder that may affect the subject's compliance with the study.
22. The subject has a pre-existing or persistent clinically significant disease, medical condition, surgical history, abnormal physical examination findings, or laboratory tests that, in the opinion of the investigator, are not in the best interest of the subject; or may alter the absorption, distribution, metabolism, or excretion of the study treatment; or impair the assessment of the study results.
23. unwillingness or inability to comply with the study procedures and study limitations or which, in the investigator's judgment, would make the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 2 years
  Number of patients with adverse events by system organ class and preferred term
Incidence of Serious Adverse Events (SAEs) | 2 years
  Number of patients with serious adverse events by system organ class and preferred term
Incidence of dose-limiting toxicities (DLT) as defined in the protocol | 2 years
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Incidence of baseline laboratory finding, ECG and vital signs changes | 2 years
  measured by laboratory and vital sign variables over time including change from
Proportion of patients with radiological response (ORR) | 2 years
  Assessed by overall response rate (ORR) defined as the proportion of patients who have a confirmed complete or partial radiological response by the Investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The percentage or number of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST v1.1)
Duration of Response (DoR) | 2 years
  The percentage of patients with confirmed CR or PR or having SD maintained (RECIST v1.1)
Disease Control Rate (DCR) | 2 years
  From date of first dose of ANS014004 up until progression, or the last evaluable assessment in the absence of progression
Progression free Survival (PFS) | 2 years
  The time from first dose until RECIST 1.1 defined disease progression or death due to any cause
Overall Survival (OS) | 2 years
  The time from the date of the first dose of study treatment until death due to any cause
Pharmacokinetics of ANS014004: Plasma PK concentrations | 2 years
  Measurement of plasma concentrations of ANS014004, total antibody and total unconjugated warhead
Pharmacokinetics of ANS014004: Area under the concentration time curve (AUC) | 2 years
  Measurement of PK parameters: Area under the concentration time curve (AUC)
Pharmacokinetics of ANS014004: Maximum plasma concentration of the study drug (C-max) | 2 years
  Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max)
Pharmacokinetics of ANS014004: Time to maximum plasma concentration of the study drug (T-max) | 2 years
  Measurement of PK parameters: Time to maximum observed plasma concentration of the study drug (T-max)
Pharmacokinetics of ANS014004: Clearance | 2 years
  Measurement of PK parameters: the volume of plasma from which the study drug is completely removed per unit time (Clearance)
Pharmacokinetics of ANS014004: Half-life | 2 years
  Measurement of PK parameters: Terminal elimination half-life (t 1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Ph.D Shun Lu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No